CLINICAL TRIAL: NCT01520272
Title: Immunogenicity of Bivalent HPV Vaccine Among Partially Vaccinated Young Adolescent Girls in Uganda
Brief Title: HPV Vaccine Effectiveness in Partially Vaccinated Girls in Uganda
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912021; 12-C-N021
Record Dates: First submitted 2012-01-26; First posted 2012-01-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-06-28

CONDITIONS: HPV16 Anitbody Levels Post Vaccination; HPV18 Antibody Levels Post Vaccination
Keywords: HPV18 Immunogenicity; HPV16 Immunogenicity; Bivalent HPV16/18 Vaccine; Less than 3 Dosed of the Bivalent HPV Vaccine; HP Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Cervical cancer is one of the leading causes of cancer death in women worldwide and in Uganda. It is caused by the human papillomavirus (HPV). A vaccine against HPV was offered for all 10-year-old girls in the Nakasongola district of Uganda from October 1, 2008, to October 31, 2009. The HPV vaccine requires three doses; however, some girls received only one or two doses. Researchers want to compare vaccine immunogenicity in girls who received all three doses with those who had only one or two doses.

Objectives:

- To examine the immunogenicity (antibody levels) of girls in Uganda who received only one, two or three doses of HPV vaccine.

Eligibility:

* Girls who will be at least 12 years old by October 31, 2011, and had at least one dose of the HPV vaccine.
* All participants will come from the Nakasongola district of Uganda.

Design:

* Participants will have a physical exam and answer questions about their medical history and HPV risk.
* Participants will provide a single blood sample for testing.
* Treatment and vaccines will not be provided as part of this study. Girls who did not receive all three doses of the HPV vaccine will be given information about the nearest health center. Health centers will provide the missed doses free of charge.

DETAILED DESCRIPTION:
Background:

Recent experience with HPV vaccine implementation in low resource settings has suggested that high vaccine coverage for all three doses could be achieved provided programs are planned well and have full and complementary components in place. However, some locations experienced substantial rates of partially vaccinated girls, those who received only one or two doses. From the vaccine trial data published thus far, we know that the vaccines produce high levels of type-specific anti-HPV antibodies which begin to stabilize past 24 months post-vaccination. Without an immune correlate of protection, it is difficult to know whether girls who received one or two vaccine doses will still experience the same benefit of protection from HPV infection as those who received all three doses of vaccine.

Recent data from a trial of a two-dose regimen of vaccination of girls aged 9-13 years in Vancouver, Canada have suggested that the immune response of girls who received only two doses was non-inferior both to that of girls who received 3 doses and to that of adult women aged 16-25 years who also received 3 doses. In a complementary study in Guanacaste, Costa Rica, vaccine efficacy (defined as 12-month vaccine type-specific infection persistence) among adult women who received either one or two doses of HPV vaccine as a part of the Phase IIb clinical trials of Cervarix (GSK) was similar to women who received all three vaccines doses.

This proposed study would provide additional insight into the immunogenicity of HPV vaccine among partially vaccinated girls in Uganda, which could add supportive evidence in an African adolescent population (currently not represented in any clinical studies of HPV vaccines) of the immunological implications of receiving less than 3 doses of HPV vaccine.

Objective:

To investigate whether the anti-HPV 16 and/or anti-HPV-18 immune responses elicited by the bivalent vaccine for girls who received one dose and those who received two doses are similar at greater than or equal to 24 months (after last dose) to girls who received all three doses of bivalent HPV vaccine.

Eligibility:

Girls who received at least one dose of the HPV vaccine, 12-20 years of old, in apparent good general health.

Design:

This is a cross-sectional immunogenicity study with three groups:

Group 1 - 200 girls who received only one dose of HPV vaccine as a part of the PATH-UNEPI HPV vaccine demonstration project;

Group 2 - 200 girls who received only two doses of HPV vaccine as a part of the PATH-UNEPI

HPV vaccine demonstration project; and

Group 3 - 200 girls who received all three doses of HPV vaccine as a part of the PATH-UNEPI HPV vaccine demonstration project.

This study will enroll girls (by group) within one district of Uganda from an HPV vaccine registry maintained by the district.

Antibody level will be parameterized as the geometric mean titre of serum antibody to HPV types 16 and/or 18 at greater than or equal to 24 months after last dose of vaccine. Titres will be measured using the polyclonal Direct VLP ELISA.

ELIGIBILITY:
* INCLUSION CRITERIA:

The following inclusion criteria will be reviewed at the time of enrollment, and where noted, confirmed at the clinic visit, immediately prior to blood draw:

* Subject is aged 12-17 years as of August 31, 2011.
* Subject received at least one dose of HPV vaccine, Cervarix (GSK, UK), from October 1, 2008 through October 31, 2009 as a part of the PATH HPV vaccine demonstration project in Nakasongola, Uganda.
* Signed and dated informed written consent form (with both parent and subject s signatures) received (confirmed at clinic visit).
* Subject is afebrile, in good apparent health (confirmed at clinic visit).
* Subject assents to participate (confirmed at clinic visit).
* Subject is able to comply with the study protocol (confirmed at clinic visit).
* Subject plans to stay in Nakasongola for the duration of enrolment, which is expected to be about week between signed consent and blood draw.

EXCLUSION CRITERIA:

The following exclusion criteria will be reviewed at the time of enrollment, and where noted, confirmed at the clinic visit.

* Prior HPV vaccination outside the PATH HPV vaccine demonstration project period.
* Subject is known to be pregnant or lactating at the time of the scheduled blood draw (confirmed at clinic visit).
* Subject has an apparent moderate or severe acute illness or has fever (confirmed at clinic visit).
* Clinical history of bleeding disorders such as haemophilia, thrombocytopenia, or anticoagulant therapy.
* Investigational drug or investigational vaccine or licensed vaccine administered during the period from 30 days before the date of the scheduled blood draw (confirmed at clinic visit).
* Subject receives immunoglobulins and/or any blood products during the period from 30 days before the date of the scheduled blood draw (confirmed at clinic visit).
* Subject or subject s parents refused to sign written consent.
* Subject does not assent at the time of the blood draw.

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 376 (Actual)
Dates: Start 2012-01-02; Study Completion 2017-06-28

PRIMARY OUTCOMES:
HPV Immunogenicity | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hildesheim, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- District of Nakasangola, Kampala, Uganda

REFERENCES:
- [Background] Banura C, Mirembe FM, Katahoire AR, Namujju PB, Mbonye AK, Wabwire FM. Epidemiology of HPV genotypes in Uganda and the role of the current preventive vaccines: A systematic review. Infect Agent Cancer. 2011 Jul 12;6(1):11. doi: 10.1186/1750-9378-6-11. PMID 21749691
- [Background] Block SL, Nolan T, Sattler C, Barr E, Giacoletti KE, Marchant CD, Castellsague X, Rusche SA, Lukac S, Bryan JT, Cavanaugh PF Jr, Reisinger KS; Protocol 016 Study Group. Comparison of the immunogenicity and reactogenicity of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in male and female adolescents and young adult women. Pediatrics. 2006 Nov;118(5):2135-45. doi: 10.1542/peds.2006-0461. PMID 17079588
- [Background] Centers for Disease Control and Prevention (CDC). National, state, and local area vaccination coverage among adolescents aged 13-17 years --- United States, 2009. MMWR Morb Mortal Wkly Rep. 2010 Aug 20;59(32):1018-23. PMID 20724968